CLINICAL TRIAL: NCT01201850
Title: The Role of Bevacizumab in the Treatment of Radiation Necrosis in Children With Central Nervous System Tumors
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Poor accrual
Sponsor: University of Colorado, Denver (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10-0418.cc
Record Dates: First submitted 2010-09-13; First posted 2010-09-15 (Estimated); Results first posted 2021-04-29 (Actual); Last update posted 2021-05-19 (Actual); Status verified 2021-04

CONDITIONS: Radiation Necrosis
Keywords: radiation necrosis; Bevacizumab (Avastin®); Central Nervous System Tumors
MeSH Terms: conditions — Central Nervous System Neoplasms | interventions — Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Bevacizumab (Avastin®) (Experimental): Once enrolled on study, patients will be treated with bevacizumab (10mg/kg) intravenously (i.v.) every 2 weeks for a total of 6 doses.
  Interventions: Drug: Bevacizumab (Avastin®)

INTERVENTIONS:
Drug: Bevacizumab (Avastin®) — Once enrolled on study, patients will be treated with bevacizumab (10mg/kg) intravenously (i.v.) every 2 weeks for a total of 6 doses. An MRI will be done after the first cycle (3 doses/ 6weeks) and then again at the end of therapy.

SUMMARY:
This study is being done to learn about the safety of the study drug bevacizumab(Avastin®), when used to treat radiation necrosis.

The primary objective of this study is to test the feasibility of treating Central Nervous System (CNS) tumor patients suffering from radiation necrosis with bevacizumab every 2 weeks.

The secondary objectives of this study are:

* To evaluate improvement in neurologic symptoms associated with bevacizumab as assessed by clinical evaluation;
* To investigate the neuro-imaging changes in radiation necrosis associated edema, including Mass Resonance (MR) spectroscopy;
* To evaluate changes in corticosteroid use in patients with radiation necrosis following treatment with bevacizumab;
* To evaluate changes in quality of life.

DETAILED DESCRIPTION:
Treatment Plan:

For patient consented and enrolled on study, bevacizumab will be administered at a dose of 10 mg/kg IV every 2 weeks for a total of 6 doses (3 doses/cycle).

Patients are expected to receive at least 1 cycle (6 weeks) of study treatment unless an unacceptable drug reaction occurs. Patients will receive a second cycle of treatment as long as treatment is tolerated. Response assessment will be performed every 6 weeks (three doses/cycle of study drug) including clinical and radiological assessment. Secondary measures including documentation of total equivalent steroid dose, length of time on steroids, and quality of life using the modified McMaster Health Instrument scale will also be collected while on treatment and 30 days after finishing treatment.

Safety will be assessed by routine physical and laboratory evaluations. Adverse events will be recorded and the severity graded according to the NCI Common Terminology Criteria for Adverse Events (version 4.0).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 1 and < 25 years of age at diagnosis
* Interval from radiation therapy at least 4 weeks and no more than 1 year
* Neurologic deterioration (long tract signs, cranial nerve signs or ataxia) consistent with radiation necrosis
* MRI imaging with findings consistent with radiation necrosis as confirmed by the study radiologist
* Craniotomy or intracranial biopsy site must be adequately healed, free of drainage or cellulitis, and the underlying cranioplasty must appear intact at the time of study entry
* More than 28 days elapsed from the last surgical procedure (including biopsy, surgical resection, wound revision, or any other major surgery involving entry into a body cavity)
* Lansky or Karnofsky performance > 40%
* Patients may be on steroids at study entry
* Adequate organ function defined as:

  * Peripheral absolute neutrophil (ANC) >/= 1000/units/Liter(uL)
  * Platelet count >/= 50,000/uL
  * Hemoglobin >/= 9.0 gm/dL (transfusion permitted)
  * Adequate Coagulation function defined as:

    * Prothrombin Time (PT)/activated Partial Thromboplastin Time (aPTT) </= 1.5x institutional upper limit of normal (ULN) for age;
  * Adequate Renal Function defined as:

    * Serum creatinine </= 1.5x institutional upper limit of normal (ULN) for age. If the serum creatinine is above these values, the calculated creatinine clearance or radioisotope Glomerular Filtration Rate (GFR) must be >/= 60 mL/min/1.73m2;
  * Adequate Hepatic Function defined as:

    * Total bilirubin </= 1.5x institutional upper limit of normal (ULN);
    * Alanine Amniotransferase (ALT) and Aspartate Aminotransferase(AST) </= 2.5x ULN for institution;Serum albumin </= 2.0 g/dL;
  * QT corrected (QTc) interval within normal range for age;
  * Adequate Pulmonary Function defined as:

    * Room air oxygen saturation of >90% at altitude > 5000 feet, or >93% < 5000 feet
* Chemotherapy: Patients must have fully recovered from the acute toxic effects of all prior chemotherapy prior to entering study. Three (3) weeks must have elapsed since the administration of prior chemotherapy.
* Biologic agents: At least 14 days must have elapsed since the completion of therapy with a monoclonal antibody
* Stem cell transplant: patients who have undergone prior stem cell transplant will not be excluded from study entry as long as adequate marrow reserve is demonstrated (refer to hematologic parameters).
* For females of childbearing potential, a negative serum pregnancy test must be documented prior to enrollment
* Patients who enter this study and their sexual partners who are of childbearing potential must agree to use an effective form of contraception throughout participation in this study
* Written informed consent and assent as required by institutional guidelines

Exclusion Criteria:

1. Disease-Specific Exclusions

   •Evidence of recent (less than 2 weeks) hemorrhage on postoperative MRI of the brain. However, patients with clinically asymptomatic presence of hemosiderin, resolving hemorrhagic changes related to surgery, and presence of punctate hemorrhage in the tumour are permitted entry into the study.
2. General Medical Exclusions

   * Subjects meeting any of the following criteria are ineligible for study entry:
   * Inability to comply with study and/or follow-up procedures
   * Life expectancy of less than 12 weeks
   * Patients who have had chemotherapy within three (3) weeks or radiation within four (4) weeks. Patients may not receive additional chemotherapeutic agents while on this study.
   * Current, recent (within 4 weeks of the first infusion of this study), or planned participation in an experimental drug study other than a Genentech-sponsored bevacizumab cancer study
   * Active second malignancy, other than superficial basal cell and superficial squamous (skin) cell, or carcinoma in situ of the cervix within last five years.
3. Bevacizumab-Specific Exclusions

   * Inadequately controlled hypertension (defined as above the normal published range for age and height)
   * Prior history of hypertensive crisis or hypertensive encephalopathy
   * New York Heart Association (NYHA) Grade II or greater congestive heart failure
   * History of myocardial infarction or unstable angina within 12 months prior to Day 1
   * No history of stroke or transient ischemic attack
   * Significant vascular disease (e.g., aortic aneurysm, requiring surgical repair or recent peripheral arterial thrombosis) within 6 months prior to Day 1; History of hemoptysis (greater than or equal to 1/2 teaspoon of bright red blood per episode) within 1 month prior to Day 1
   * Evidence of bleeding diathesis or significant coagulopathy (in the absence of therapeutic anticoagulation)
   * Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to Day 1 or anticipation of need for major surgical procedure during the course of the study
   * Core biopsy or other minor surgical procedure, excluding placement of a vascular access device, within 7 days prior to Day 1
   * History of abdominal fistula or gastrointestinal perforation within 6 months prior to Day 1
   * Serious, non-healing wound, active ulcer, or unhealed bone fracture
   * Proteinuria as demonstrated by a Urine Protein Creatinine (UPC) ratio greater than or equal to 1.0 at screening
   * Known hypersensitivity to any component of bevacizumab
   * Pregnancy (positive pregnancy test) or lactation. Use of effective means of contraception (men and women) in subjects of child-bearing potential

Ages: 1 Year to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 7 (Actual)
Dates: Start 2010-06-28 (Actual); Primary Completion 2016-08-04 (Actual); Study Completion 2016-08-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Margaret Macy, MD, Principal Investigator — Children's Hospital Colorado
Locations (1):
- Children's Hospital Colorado, Aurora, Colorado, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Bevacizumab (Avastin®): Once enrolled, patients were treated with bevacizumab (10mg/kg) intravenously (i.v.) every 2 weeks for a total of 6 doses.
  Bevacizumab (Avastin®): bevacizumab (10mg/kg) intravenously (i.v.) every 2 weeks for a total of 6 doses.
Period: Overall Study
Arm/Group | Bevacizumab (Avastin®)
Started | 7
Completed | 3
Not Completed | 4
Not completed — Tumor progression | 4

BASELINE CHARACTERISTICS:
Arm/Group | Bevacizumab (Avastin®)
Number analyzed (Participants) | 7
Age, Customized [Number; unit: participants]
  <10 yrs | 3
  >10 and <26 yrs | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 5
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Received at Least 5 of the 6 Scheduled Doses of Bevacizumab
Description: This pilot study was designed to evaluate the feasibility of treating pediatric patients with CNS radiation necrosis with bevacizumab. Patients enrolled on study were assessed for number of doses of bevacizumab that they received while on study. Participants who successfully received at least 5 of the 6 planned doses of bevacizumab (IV every 2 weeks) without significant events were determined to have met the outcome measure.
Time Frame: 13 weeks
Population: All patients who were enrolled/received a dose of bevacizumab were assessed.
Measure: Number; unit: participants
Arm/Group | Bevacizumab (Avastin®)
Number analyzed (Participants) | 7
participants | 3

2. Secondary Outcome: Neurologic Status With Bevacizumab Treatment
Description: Outcome 1: Monitor overall neurologic status and symptoms before, during and 1 month following treatment with bevacizumab.
Time Frame: 13 weeks
Population: Monitor overall neurologic status and symptoms before, during and 1 month following treatment with bevacizumab.
Measure: Number; unit: participants
Arm/Group | Bevacizumab (Avastin®)
Number analyzed (Participants) | 7
participants
  Neurologic improvement | 4
  No Neurologic improvement | 3

3. Secondary Outcome: Corticosteroid Usage With Bevacixumab Treatment
Description: Outcome 2: Dose and duration of corticosteroid use prior to, during, and up to 1 month following bevacizumab treatment will also be collected and evaluated.
Time Frame: 13 weeks
Population: The dose and duration of corticosteroid use was collected and evaluated.
Measure: Mean (Standard Deviation); unit: milligram
Arm/Group | Bevacizumab (Avastin®)
Number analyzed (Participants) | 7
milligram
  Baseline Dexamethasone Dose (mg) | 6.0 (4.0)
  End of therapy Dexamethasone dose (mg) | 2.3 (5.2)

4. Secondary Outcome: Changes in Quality of Life With Bevacizumab Treatment
Description: Outcome 3: To evaluate changes in quality of life before and after treatment with bevacizumab Modified McMasters Scale was used. Minimum score: 1 Maximum score 35. Higher score indicates worse quality of life.
Time Frame: 13 weeks
Population: The participant's quality of life as determined by the Modified McMaster Scale was evaluated at baseline, during and after treatment with bevacizumab
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Bevacizumab (Avastin®)
Number analyzed (Participants) | 7
score on a scale
  Baseline Modified McMasters Score | 14.4 (3.6)
  End of therapy Modified McMasters Score | 15.3 (4.5)

5. Secondary Outcome: Number of Patients With Changes in Neuro-Imaging With Bevacizumab Treatment
Description: Outcome 4: To investigate the neuro-imaging changes in radiation necrosis associated edema, including Mass Resonance (MR) spectroscopy; MRIs (including FLAIR sequences and contrast enhanced images) were evaluated for changes in the radiation necrosis imaging characteristics by a pediatric radiologist. Decreases in gadolinium enhancement, FLAIR signal were considered changes consistent with decreased edema. Tumor size was also evaluated, with a decrease in tumor size indicating decreased edema/improved radiation necrosis
Time Frame: 13 weeks
Population: Descriptive report of radiographic changes with bevacizumab treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Bevacizumab (Avastin®)
Number analyzed (Participants) | 7
Participants
  Decreased gadolinium enhancement | 7
  Decreased FLAIR signal | 5
  Decreased tumor size | 5

ADVERSE EVENTS:
Time Frame: 16 weeks (duration of trial and 30 days post last dose of bevacizumab)
Description: Adverse events that were possibly, probably or definitely related to study therapy were reported.
Arm/Group | Bevacizumab (Avastin®)
All-Cause Mortality (participants affected / at risk) | 0/7
Serious Adverse Events (participants affected / at risk) | 0/7
Other Adverse Events (participants affected / at risk) | 4/7
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Bevacizumab (Avastin®) (N=7)
Aspartate aminotransferase increased (Investigations) | 1
epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
proteinuria (Renal and urinary disorders) | 2
renal and urinary disorders, other (Renal and urinary disorders) | 1 — dysuria
back pain (Musculoskeletal and connective tissue disorders) | 1
mucositis (Gastrointestinal disorders) | 1
lymphocyte count decreased (Investigations) | 2
hypophosphatemia (Investigations) | 1
hypomagnesemia (Investigations) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No